CLINICAL TRIAL: NCT07307261
Title: Evaluation of Mirabegron Versus Tamsulosin or Their Combination in Treatment of Lower Urinary Tract Symptoms Related to Double j Stent in Adults: A Prospective Randomized Study
Brief Title: Evaluation of Mirabegron Versus Tamsulosin or Their Combination in Treatment of Lower Urinary Tract Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avraiem Talaat (Other)
Responsible Party: Sponsor-Investigator, Avraiem Talaat, Resident at Urology Department, South Valley University
Organization: South Valley University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mirabegron Vs Tamsulosin
Record Dates: First submitted 2025-01-19; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2024-10

CONDITIONS: Ureteric Stent-related Morbidity
MeSH Terms: interventions — Tamsulosin; mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tamsulosin 0.4mg (Active Comparator): About 100 patients will receive Tamsulosin (0.4mg) once daily for 3 weeks for the treatment of lower urinary tract symptoms related to double j stent in adults
  Interventions: Drug: Tamsulosin
- Mirabegron 50mg (Active Comparator): About 100 patients will receive Mirabegron (50mg) once daily for 3 weeks for the treatment of lower urinary tract symptoms related to double j stent in adults
  Interventions: Drug: Tamsulosin
- combination of tamsulosin 0.4mg and Mirabegron 50mg (Active Comparator): About 100 patients will receive A combination of tamsulosin (0.4mg) and Mirabegron (50mg) once daily for 3 weeks for the treatment of lower urinary tract symptoms related to double j stent in adults
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Tamsulosin — to compare the effect of mirabegron and tamsulosin and their combination on ureteric stent-related morbidity
  Other Names: Mirabegron

SUMMARY:
Stent related symptoms (SRSs) comprise of complaints such as irritative symptoms, sense of incomplete emptying, flank and suprapubic pain, and incontinence. Mechanical irritation of trigone, urinary reflux, and stent movement are plausible causes for SRSs.

Alpha-blockers are the primary medications for ureteral stent-related symptoms. These medications are suggested to patients by the American Urological Association (AUA)/Endourological Society guideline to reduce stent-related symptoms with moderate recommendation. Nevertheless, there are many side effects associated with alpha-blockers such as dizziness, headache, and orthostatic hypotension

DETAILED DESCRIPTION:
Ureteral stents have become an important part of urologic practice since first described the double-J stent . most often urolithiasis. Their use may be associated with significant bothersome symptoms and discomfort. Ureteral stent-related symptoms (SRSs) may occur in up to 88% of patients in mild or more severe degree.

Mirabegron is the first and only selective β3-adrenergic receptor agonist agent currently available and it is one of the treatment options for overactive bladder (OAB). Hence, many urologists have been introducing mirabegron therapy for OAB in recent years and because the SRS are similar to OAB symptoms, it may be another treatment option for reducing bladder irritability in patients indwelling DJ stent.

It is currently unclear whether mirabegron has a place in the treatment of SRSs. Our study aims to systematically evaluate the efficacy and safety of mirabegron in treating SRSs in comparison to Tamsulosin and their combination in adult patients

ELIGIBILITY:
Inclusion Criteria:

* First time to use Ureteric stent .

Exclusion Criteria:

* Urinary tract infection.
* Previous ureteral surgery.
* Congenital malformation of the ureter.
* Distal ureteric stricture.
* Hypersensitivity to the drugs.
* Pregnancy or lactation.
* Hepatic insufficiency
* Non-compliant patients.
* Age < 18 years old .

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-10-05 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Treatment of Ureteral Stent Pain | 4 Weeks
  All patients will be evaluated before and after the treatment from the pain by the visual analog pain scale..

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Sayed Abdel-kader, Professor, Study Chair — Urology Department,faculty of Medicine, South Valley university.
Locations (1):
- Qena Hospital, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Undecided